CLINICAL TRIAL: NCT02179060
Title: Prehospital Resuscitation Intranasal Cooling Effects Seen in Magnetic Resonance Imaging of the Brain After Cardiac Arrest
Brief Title: Prehospital Resuscitation Intranasal Cooling Effects Seen in MRI of the Brain After Cardiac Arrest
Acronym: COOLCAMRI
Status: Terminated | Type: Observational
Why Stopped: Lack of study funding
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Helsinki University Central Hospital (Other); BeneChill, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: R14025
Record Dates: First submitted 2014-06-02; First posted 2014-07-01 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Arrest
Keywords: Sudden cardiac arrest, RhinoChill -cooling, MRI
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cooling group: The RhinoChill® cooling is started as soon as possible to the patients with Cardiac arrest, and before the return of spontaneous circulation
- Control group: Standard care, no cooling during pre-hospital care

SUMMARY:
Therapeutic hypothermia improves the neurologically-intact survival rates in those patients resuscitated out-of-hospital from ventricular fibrillation. Cooling as early as possible might be beneficial to those victims. Diffusion Tensor Imaging and diffusion-weighted magnetic resonance imaging have recently shown to be able to identify early ischemia-related changes within the brain three days after cardiac arrest, among sudden cardiac arrest patients cooled in hospital. The physical changes seen within the brain may be able to distinguish survivors at very early phase.

This study aims to assess early ischemia-related changes of the brain seen in MRI approximately three days after cardiac arrest. The hypotheses is that MRI will differ in the groups of patients treated with early intra-arrest cooling with the RhinoChill device and in hospital hypothermia in 36 Celsius, in the group of patients treated with normal in hospital hypothermia in 36 Celsius only, in the group of patients treated with normal in hospital hypothermia in 33 Celsius only (The historical Xenon study patients). The primary endpoint is the presence and pattern of white matter and gray matter degeneration and volumetric changes of the gray matter, white matter, and cerebro-spinal fluid spaces in MRI, and secondary endpoints are total survival at 90 days, and time to reach a target temperature (≤36/33 Celsius).

DETAILED DESCRIPTION:
Medical personnel (e.g,. nurses or physicians) responding to a cardiac arrest will assess each patient for study inclusion. During resuscitation patients will receive standard ALS (advanced life support) according to European Resuscitation Council (ERC) guidelines with cooling with the RhinoChill upon determining that the patient is in cardiac arrest. The RhinoChill catheters should be placed and cooling initiated immediately after airway management (i.e. laryngeal mask or intubation). The aim is that cooling should be started within 15 minutes from the call to the dispatch centre. Specifically, cooling with chilled saline or cold packs in the field or ambulance will not be permitted. Resuscitation attempts should be continued for at least 45 minutes after the collapse in all patients having venticular fibrillation (VF) or non-perfusive venticular tachycardia (VT) as initial cardiac rhythm before deciding that further interventions are futile.

Automated external defibrillator (AEDs) with the capability to record data will be used in each resuscitation attempt, and the quality of cardio pulmonary resuscitation (CPR) is followed.

RhinoChill cooling will be continued in those subjects that achieve ROSC and remain comatose. Bolus doses of sedation and analgesia will be administered for their transport to the hospital according to local protocol. RhinoChill cooling will be continued at the hospital until the subject can be successfully transitioned to the standard institutional cooling protocol.

Clinical assessments and clinically relevant adverse events will be documented from the time the patient is enrolled to the study until the first of the following two events occur: death or MRI scan.

Patients that regain consciousness following ROSC and prior to hospital transport will be excluded. Patient's still unconscious in the emergency room are admitted to ICU and therapeutic cooling is continued for 24 to 36 hours. The MRI scan will take place within 16 hours after rewarming. After that the sedation is stopped and patient extubated if possible. The study is finished at that point and normal patient care continues.

The study continues until 10 patients with MRI scan are enrolled in Tampere University Hospital (TAUH).

ELIGIBILITY:
Inclusion Criteria:

1. Ventricular fibrillation or non-perfusive ventricular tachycardia as initial cardiac rhythm.
2. The 1st attempt at resuscitation by emergency medical personnel must appear within 15 minutes after the collapse.
3. The cause for collapse should be considered primary as cardiogenic and the return of spontaneous circulation (ROSC) should have been gained in 45 minutes after the collapse.
4. Patient should be still unconscious in the emergency room.
5. Age: 18 - 80 years
6. Obtained consent after arrival to the hospital, and before MRI scan.

   Exclusion Criteria:
7. Hypothermia (< 30°C core temperature)
8. Arrival of EMS after 15 minutes from collapse
9. Unconsciousness before cardiac arrest (cerebral trauma, spontaneous cerebral haemorrhages, intoxications etc.)
10. Terminal phase of a chronic disease, or known limitations in therapy and Do Not Resuscitate-order or known pre-arrest Cerebral Performance Category 3 or 4
11. Factors making participation in follow-up unlikely
12. Factors making the RhinoChill cooling contraindicated: patients with known contraindications to hypothermia (Raynaud's disease, Cryoglobulinemia, Sickle Cell disease), have specific temperature-sensitive pathologies (e.g., serum cold agglutinins, Buerger's disease), intranasal obstruction, or known skull base fracture.
13. Pregnancy
14. Coagulopathy
15. Response to verbal commands after the return of spontaneous circulation (ROSC)
16. Systolic arterial pressure < 80 mmHg or mean arterial pressure < 60 mmHg for over 30 min period after ROSC
17. Evidence of hypoxemia (arterial oxygen saturation < 85%) for > 15 minutes after ROSC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be derived from the prehospital cardiac arrest patients from Tampere area treated by the Tampere Area Emergency Medical Service (EMS) led by physician. The study population (N=10) is from Pirkanmaa area. The paramedics are allowed to start intra-arrest cooling by RhinoChill whenever they meet an adult SCA patient in VF/VT. The third group of control subjects are same as used in "Effect of Xenon, in Combination with Therapeutic Hypothermia, on the Brain and on Neurological Outcome following Brain Ischemia in Cardiac Arrest Patients (EudraCT number 2009-009505-25)" -study running in Turku and Helsinki, Finland. They are the prehospital cardiac arrest patients from Turku and Helsinki area treated by the Turku or Helsinki Area Emergency Medical Service.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
the presence and pattern of white matter and gray matter degeneration and volumetric changes of the gray matter, white matter, and cerebro-spinal fluid spaces in MRI | 36-49 hours after cardiac arrest

SECONDARY OUTCOMES:
the total survival at 90 days | 90 days after cardiac arrest

OTHER OUTCOMES:
time to reach a target temperature (≤36/33 Celsius) | 0-12hours after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Hoppu, MD, PhD, Principal Investigator
Locations (1):
- Tampere University hospital, Tampere, Finland